CLINICAL TRIAL: NCT05946434
Title: Comparisons of the Effects of Kinesio Taping and Rigid Taping in Knee Osteoarthritis
Brief Title: Effects of KT and Rigid Taping in Knee OA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Muhammad Saad
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis, kinesio tape and rigid tape
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Tape Group (Experimental): Kinesio tape applied along with conventional treatment
  Interventions: Other: Kinesio Tape Group; Other: Rigid Tape Group
- Rigid tape Group (Experimental): Rigid tape applied along with conventional treatment
  Interventions: Other: Kinesio Tape Group; Other: Rigid Tape Group

INTERVENTIONS:
Other: Kinesio Tape Group — Physiotherapy Protocol Followed:
  * Hot pack and TENS application for 10 minutes.
  * Knee isometric exercises by placing roller beneath knee joint and pressing it by keeping leg straight and holding it for 10-15 seconds with 10 repetitions.
  * Stretching of hamstrings and gastrocnemius muscles, maintaining stretch for 20 seconds and 7 repetitions should be performed.
  * Tibio-femoral glides and patellar mobilizations will be performed.
  * At the end kinesio taping will be performed at knee joint for inhibition.
  Same procedure will be followed in all follow ups at day 1, day 14 and day 28.
Other: Rigid Tape Group — Physiotherapy Protocol Followed:
  * Hot pack and TENS application for 10 minutes.
  * Knee isometric exercises by placing roller beneath knee joint and pressing it by keeping leg straight and holding it for 10-15 seconds with 10 repetitions.
  * Stretching of hamstrings and gastrocnemius muscles, maintaining stretch for 20 seconds and 7 repetitions should be performed.
  * Tibio-femoral glides and patellar mobilizations will be performed.
  * At the end rigid tape will be applied on knee joint to provide stability.
  Same procedure will be followed in all follow ups at day 1, day 14 and day 28

SUMMARY:
The purpose of the study is to compare the effects of kinesio taping and rigid taping in Knee Osteoarthritis to alleviate symptoms like pain, reduce range of motion and functional limitations. A randomized control trial was conducted at Atta Memorial Hospital, Airport Society, Rawalpindi and Makkah Medical Complex, Rawalpindi. The sample size was 36 calculated through G-Power. The participants were divided into two interventional groups each having 18 participants. The study duration was six months. Sampling technique applied was Non probability convenient sampling. Only 40 to 60 years' participants with grade 1-3 Knee Osteoarthritis according to kellgren-Lawrence scale were included in the study. Tools used in this study are Visual analogue scale, WOMAC Index, timed up and go test and Goniometer self-structured Questionnaire. Data was collected before and immediately after the application of intervention on First day and then again at the end of session on 14th and 28th day. Data analyzed through SPSS version 23.

DETAILED DESCRIPTION:
Osteoarthritis (OA), also referred to as degenerative joint disease, primary OA, wear-and-tear arthritis, or age-related arthritis, is the most common cause of disability in the US and around the world. In medical terminology, arthritis refers to joint inflammation. More than 100 rheumatic diseases and ailments that affect the joints, the tissues surrounding the joints, and other connective tissue are collectively referred to as arthritis in the public health sector(1). By 2020, OA will rank as the fourth most common cause of disability, according to the World Health Organization (WHO), making it one of the most incapacitating musculoskeletal ailments. Globally, the socioeconomic, psychological, and physical toll increased. The main leading factor affecting mobility is knee osteoarthritis. Among patients with knee OA, knee discomfort, decreased knee flexibility, and functional impossibility are frequent clinical symptoms during daily activities(2). Almost any joint can be compromised by osteoarthritis, although the hands, knees, hips, and feet are the most frequently affected ,but most commonly involved joint is knee joint(3). Knee osteoarthritis (OA) is a prevalent, degenerative, multifactorial joint condition that is characterized by chronic pain and functional dysfunction . Nearly half of all OA cases worldwide are knee OA, which gets worse as people get older and more obese(4, 5). Knee discomfort, which contributes to OA, was also brought on by inactivity or a sedentary lifestyle. In order to prevent pain when engaging in physical activity, people with knee OA further restrict their mobility(6).

Diagnosis of Knee Osteoarthritis: The presence of typical symptoms, physical exam findings, test data, and imaging characteristics all help to confirm a medical diagnosis of knee OA. Knee osteoarthritis can't be diagnosed based on single finding from the followings Literature review: The randomized control trial was conducted in Turkey on osteoarthritis patient to see the effect of kinesio taping results indicate that there were clear decrease in Nottingham Health Profile (NHP) scores (15). In this study there were 13 males (32%) and 28 females (68%). In both groups (K Tape and sham tape) VAS for activity pain, VAS for nocturnal pain, Lequesne index score, NHP score decreased significantly. NHP energy scores were different significantly between the groups in favor of sham taping at the end of the 12-day period. Another research conducted in Germany, the main finding of this study is that wearing a kinesio tape over 3 consecutive days is effective to improve the self-reported perception of pain, joint stiffness, and physical function in patients with OA compared with a sham tape or no intervention (16). The research conducted in Iran on effect of kinesio taping on functional disability in knee osteoarthritic patients result shows that in the kinesio tape group, a statistically significant improvement was observed in the reconstruction of the joint sense position at 30 and 60 angles of knee flexion before and after treatment (17). Therapeutic taping seemed to be superior to control taping in pain control for knee osteoarthritis. Non-elastic taping, but not elastic taping, provides benefits in pain reduction and functional performance (18)

ELIGIBILITY:
Inclusion Criteria:

1. Age group 40 to 60 years of age.
2. Both genders.
3. Radiological findings showing symptomatic 1-3 grade knee osteoarthritis.
4. Sub-acute and chronic knee pain.

Exclusion Criteria:

1. Systemic rheumatoid disease.
2. Hypersensitive skin or lesions in the areas of application for tapes.
3. Inability to perform functional tests needed according to the research protocol
4. Diagnosed or suspected cancer in the region.
5. Within 6 months of intra-articular injections.
6. Constant use of painkillers for alleviation of pain in different regions of the body.
7. Constant use of any orthotics.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) Osteoarthritis (OA) Index | 6 months
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis (OA) Index is a tested questionnaire to assess symptoms and physical functional disability in patients with OA of the knee and the hip

SECONDARY OUTCOMES:
ROM | 6 months.
  The Goniometer is an accurate and trustworthy way of measuring knee ROM, as well as a handy and readily available measure of outcome for scientific studies and physiotherapy practice.
Visual Analogue Scale | 6 months.
  The Visual Analogue Scale (VAS) is a pain outcome measure that is dependable, legitimate, receptive and widely utilized. It's made up of a single 10 cm horizontal line with two designations, "no pain" and "worst possible pain," positioned at each end of the line. Participants are instructed to put a pointy marker on the line representing their level of pain.
  Visual Analogue Scale has high reliability for pain which is 0.97 and has minimal measurement error which is 0.03

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScNMPT, Principal Investigator — Riphah International University
Locations (1):
- Atta Memorial Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- [Background] Melese H, Alamer A, Hailu Temesgen M, Nigussie F. Effectiveness of Kinesio Taping on the Management of Knee Osteoarthritis: A Systematic Review of Randomized Controlled Trials. J Pain Res. 2020 May 28;13:1267-1276. doi: 10.2147/JPR.S249567. eCollection 2020. PMID 32547187
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Malik FB, Memon AG, Shah S, Latif D, Afzal MF, Memon SAJTRJ. PREVALENCE OF KNEE OSTEOARTHRITIS AND QUALITY OF LIFE AMONG MIDDLE AGED ADULTS OF PAKISTAN: soi: 21-2017/re-trjvol06iss01p280. 2022;6(01):280-3.
- [Background] Sanchez C, Pesesse L, Gabay O, Delcour JP, Msika P, Baudouin C, Henrotin YE. Regulation of subchondral bone osteoblast metabolism by cyclic compression. Arthritis Rheum. 2012 Apr;64(4):1193-203. doi: 10.1002/art.33445. Epub 2011 Oct 27. PMID 22034083
- [Background] Gibson T, Hameed K, Kadir M, Sultana S, Fatima Z, Syed A. Knee pain amongst the poor and affluent in Pakistan. Br J Rheumatol. 1996 Feb;35(2):146-9. doi: 10.1093/rheumatology/35.2.146. PMID 8612027
- [Background] Ho-Pham LT, Lai TQ, Mai LD, Doan MC, Pham HN, Nguyen TV. Prevalence of radiographic osteoarthritis of the knee and its relationship to self-reported pain. PLoS One. 2014 Apr 10;9(4):e94563. doi: 10.1371/journal.pone.0094563. eCollection 2014. PMID 24722559
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Cho HY, Kim EH, Kim J, Yoon YW. Kinesio taping improves pain, range of motion, and proprioception in older patients with knee osteoarthritis: a randomized controlled trial. Am J Phys Med Rehabil. 2015 Mar;94(3):192-200. doi: 10.1097/PHM.0000000000000148. PMID 25706053
- [Background] Abulhasan JF, Grey MJJJoFM, kinesiology. Anatomy and physiology of knee stability. 2017;2(4):34.
- [Background] Masouros S, Bull A, Amis AJO, Trauma. (i) Biomechanics of the knee joint. 2010;24(2):84-91.
- [Background] Eaton CB. Obesity as a risk factor for osteoarthritis: mechanical versus metabolic. Med Health R I. 2004 Jul;87(7):201-4. PMID 15354794
- [Background] Felson DT, Lawrence RC, Dieppe PA, Hirsch R, Helmick CG, Jordan JM, Kington RS, Lane NE, Nevitt MC, Zhang Y, Sowers M, McAlindon T, Spector TD, Poole AR, Yanovski SZ, Ateshian G, Sharma L, Buckwalter JA, Brandt KD, Fries JF. Osteoarthritis: new insights. Part 1: the disease and its risk factors. Ann Intern Med. 2000 Oct 17;133(8):635-46. doi: 10.7326/0003-4819-133-8-200010170-00016. PMID 11033593
- [Background] Luijkx T, Pai VJDnahroak-a-l-f-c-o-o-o-kDp. Kellgren and Lawrence system for classification of osteoarthritis of knee. 2016;7(6).
- [Background] Sharma L. Osteoarthritis of the Knee. N Engl J Med. 2021 Jan 7;384(1):51-59. doi: 10.1056/NEJMcp1903768. No abstract available. PMID 33406330
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Zeng C, Dubreuil M, LaRochelle MR, Lu N, Wei J, Choi HK, Lei G, Zhang Y. Association of Tramadol With All-Cause Mortality Among Patients With Osteoarthritis. JAMA. 2019 Mar 12;321(10):969-982. doi: 10.1001/jama.2019.1347. PMID 30860559
- [Background] Deyle GD, Allen CS, Allison SC, Gill NW, Hando BR, Petersen EJ, Dusenberry DI, Rhon DI. Physical Therapy versus Glucocorticoid Injection for Osteoarthritis of the Knee. N Engl J Med. 2020 Apr 9;382(15):1420-1429. doi: 10.1056/NEJMoa1905877. PMID 32268027
- [Background] McAlindon TE, LaValley MP, Harvey WF, Price LL, Driban JB, Zhang M, Ward RJ. Effect of Intra-articular Triamcinolone vs Saline on Knee Cartilage Volume and Pain in Patients With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1967-1975. doi: 10.1001/jama.2017.5283. PMID 28510679
- [Background] Thorlund JB, Juhl CB, Roos EM, Lohmander LS. Arthroscopic surgery for degenerative knee: systematic review and meta-analysis of benefits and harms. BMJ. 2015 Jun 16;350:h2747. doi: 10.1136/bmj.h2747. PMID 26080045
- [Background] Shan L, Shan B, Suzuki A, Nouh F, Saxena A. Intermediate and long-term quality of life after total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Am. 2015 Jan 21;97(2):156-68. doi: 10.2106/JBJS.M.00372. PMID 25609443
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2015 Jan 9;1(1):CD004376. doi: 10.1002/14651858.CD004376.pub3. PMID 25569281
- [Background] Wang C, Schmid CH, Iversen MD, Harvey WF, Fielding RA, Driban JB, Price LL, Wong JB, Reid KF, Rones R, McAlindon T. Comparative Effectiveness of Tai Chi Versus Physical Therapy for Knee Osteoarthritis: A Randomized Trial. Ann Intern Med. 2016 Jul 19;165(2):77-86. doi: 10.7326/M15-2143. Epub 2016 May 17. PMID 27183035
- [Background] Messier SP, Mihalko SL, Legault C, Miller GD, Nicklas BJ, DeVita P, Beavers DP, Hunter DJ, Lyles MF, Eckstein F, Williamson JD, Carr JJ, Guermazi A, Loeser RF. Effects of intensive diet and exercise on knee joint loads, inflammation, and clinical outcomes among overweight and obese adults with knee osteoarthritis: the IDEA randomized clinical trial. JAMA. 2013 Sep 25;310(12):1263-73. doi: 10.1001/jama.2013.277669. PMID 24065013
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Peter WF, Jansen MJ, Hurkmans EJ, Bloo H, Dekker J, Dilling RG, Hilberdink W, Kersten-Smit C, de Rooij M, Veenhof C, Vermeulen HM, de Vos RJ, Schoones JW, Vliet Vlieland TP; Guideline Steering Committee - Hip and Knee Osteoarthritis. Physiotherapy in hip and knee osteoarthritis: development of a practice guideline concerning initial assessment, treatment and evaluation. Acta Reumatol Port. 2011 Jul-Sep;36(3):268-81. PMID 22113602
- [Background] Kocyigit F, Turkmen MB, Acar M, Guldane N, Kose T, Kuyucu E, Erdil M. Kinesio taping or sham taping in knee osteoarthritis? A randomized, double-blind, sham-controlled trial. Complement Ther Clin Pract. 2015 Nov;21(4):262-7. doi: 10.1016/j.ctcp.2015.10.001. Epub 2015 Oct 9. PMID 26573453
- [Background] Rahlf AL, Braumann KM, Zech A. Kinesio Taping Improves Perceptions of Pain and Function of Patients With Knee Osteoarthritis: A Randomized, Controlled Trial. J Sport Rehabil. 2019 Jul 1;28(5):481-487. doi: 10.1123/jsr.2017-0306. Epub 2018 Dec 12. PMID 29466081
- [Background] Yoshida A, Kahanov L. The effect of kinesio taping on lower trunk range of motions. Res Sports Med. 2007 Apr-Jun;15(2):103-12. doi: 10.1080/15438620701405206. PMID 17578750
- [Background] Ouyang JH, Chang KH, Hsu WY, Cho YT, Liou TH, Lin YN. Non-elastic taping, but not elastic taping, provides benefits for patients with knee osteoarthritis: systemic review and meta-analysis. Clin Rehabil. 2018 Jan;32(1):3-17. doi: 10.1177/0269215517717307. Epub 2017 Jun 29. PMID 28660785
- [Background] Wieczorek M, Rotonda C, Coste J, Pouchot J, Saraux A, Guillemin F, Rat AC. Trajectory analysis combining pain and physical function in individuals with knee and hip osteoarthritis: results from the French KHOALA cohort. Rheumatology (Oxford). 2020 Nov 1;59(11):3488-3498. doi: 10.1093/rheumatology/keaa148. PMID 32375174
- [Background] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Salaffi F, Leardini G, Canesi B, Mannoni A, Fioravanti A, Caporali R, Lapadula G, Punzi L; GOnorthrosis and Quality Of Life Assessment (GOQOLA). Reliability and validity of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index in Italian patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2003 Aug;11(8):551-60. doi: 10.1016/s1063-4584(03)00089-x. PMID 12880577
- [Background] Epskamp S, Dibley H, Ray E, Bond N, White J, Wilkinson A, et al. Range of motion as an outcome measure for knee osteoarthritis interventions in clinical trials: an integrated review. Physical Therapy Reviews. 2020;25(5-6):462-81.
- [Background] Hinman RS, Bennell KL, Crossley KM, McConnell J. Immediate effects of adhesive tape on pain and disability in individuals with knee osteoarthritis. Rheumatology (Oxford). 2003 Jul;42(7):865-9. doi: 10.1093/rheumatology/keg233. Epub 2003 Mar 31. PMID 12730546